CLINICAL TRIAL: NCT04509219
Title: Methylprednisolone Pulse Therapy for Coronary Artery Dilatation or Aneurysm Formation in Kawasaki Disease
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MP pulse in KD
Record Dates: First submitted 2020-07-14; First posted 2020-08-11 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-05

CONDITIONS: Mucocutaneous Lymph Node Syndrome
Keywords: Kawasaki Disease; aneurysm formation; coronary artery dilatation; Methylprednisolone; Pulse therapy
MeSH Terms: conditions — Mucocutaneous Lymph Node Syndrome; Coronary Aneurysm | interventions — Methylprednisolone

STUDY DESIGN:
Intervention Model Description: single arm, phase 1 study of methylprednisolone pulse therapy safety in treatment of aneurysm or coronary artery dilation of Kawasaki disease.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Participants treated with MP pulse (Experimental): Selected participants will be given MP pulse treatment
  Interventions: Drug: Methylprednisolone Injection

INTERVENTIONS:
Drug: Methylprednisolone Injection — methylprednisolone pulse therapy, 30mg/kg, with maximal dose of 1000mg/day, for continue 3 days.
  Other Names: methylprednisolone pulse therapy

SUMMARY:
In this study, the investigator plan to prescribe Methylprednisolone pulse therapy in Kawasaki disease patients with coronary artery lesions or aneurysm formation beyond acute stage to investigate the role for vasculitis of KD or regression of dilatation.

DETAILED DESCRIPTION:
Kawasaki disease is the most common systemic vasculitis in children. Coronary artery aneurysms may develop in 20-25% of untreated patients. Intravenous immune globulin (IVIG) can reduce coronary-artery aneurysms to 3-5%. Numerous studies and clinical trials had pointed out that corticosteroid treatment (pulse therapy or not) could lower the incidence of coronary artery abnormality in high-risk KD patients. However, the therapeutic effect of corticosteroid in KD patients with aneurysm formation after acute stage was never mentioned. There is no effective treatment for aneurysm formation available in KD after acute stage. Methylprednisolone pulse therapy (MP pulse) was used for treatment of KD during acute stage since more than 20 years ago. MP pulse plus IVIG seems not benefit for KD patients but benefit for IVIG resistant KD patients or for high-risk group of CAL formation/ IVIG resistance group. MP pulse therapy is well document used in autoimmune disease vasculitis such as SLE, rheumatoid arthritis, dermatomyosis...etc. Taking together, MP pulse is effective and safe for KD patients during acute stage. In this study, the investigators plan to use MP pulse in KD patients with CAL or aneurysm formation beyond acute stage to investigate the role of vasculitis of KD or regression of dilatation.

Methods: The investigators conducted a prospective study of methylprednisolone pulse therapy (MP pulse) for KD patients with coronary aneurysm or dilatation formation. The investigators will enroll these patients to receive methylprednisolone pulse (MP pulse, 30mg/kg, Max:1g/day for continue 3 days) for treatment. Together with other anti-inflammatory oral medicine including monteleukast, Dextromethorphan(DXM), prednisolone, and ketotifen as supplementary treatment.

The specific aim of this study is the regression of coronary artery aneurysm after MP pulse therapy.

Under the hypothesis and specific aim, the investigators plan to do in the following 3 years:

1. During the 1st year, the investigators will enroll for 5-10 cases for safety surveys including blood pressure monitoring, inflammatory markers, liver function, renal function, electrolyte imbalance, growth problems as Phase I study.
2. In the 2nd and 3rd year of this study, the investigators will enroll for 20-30 cases for an effective survey as Phase II study.

Results from this study will help clinicians to treat aneurysm formation or coronary artery dilatation in KD patients and reduce the activity limitation of patients, reduce the medical resource in those patients. The investigators may provide the first treatment for aneurysm in KD.

ELIGIBILITY:
Inclusion Criteria:

* Kawasaki disease patients with coronary artery dilation or aneurysm formation after acute stage (at lease 3 weeks after IVIG treatment)

Exclusion Criteria:

* patients meet the contraindications of Methylprednisolone sodium succinate, e.g., allergic to Methylprednisolone sodium succinate, premature infant, immune system related thrombocytopathy, immunodeficiency, any congenital diseases.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2020-04-15 (Actual); Primary Completion 2021-04-15 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events and physical effects of Methylprednisolone pulse therapy in Kawasaki disease patients with coronary artery aneurysms | 4 weeks from enrollment
  Measurement of body weight in Kilogram
Incidence of Treatment-Emergent Adverse Events and physical effects of Methylprednisolone pulse therapy in Kawasaki disease patients with coronary artery aneurysms | 8 weeks from enrollment
  Measurement of body weight in Kilogram
Incidence of Treatment-Emergent Adverse Events and physical effects of Methylprednisolone pulse therapy in Kawasaki disease patients with coronary artery aneurysms | 12 weeks from enrollment
  Measurement of body weight in Kilogram
Incidence of Treatment-Emergent Adverse Events and physical effects of Methylprednisolone pulse therapy in Kawasaki disease patients with coronary artery aneurysms | 16 weeks from enrollment
  Measurement of body weight in Kilogram
Incidence of Treatment-Emergent Adverse Events and physical effects of Methylprednisolone pulse therapy in Kawasaki disease patients with coronary artery aneurysms | 20 weeks from enrollment
  Measurement of body weight in Kilogram
Incidence of Treatment-Emergent Adverse Events and physical effects of Methylprednisolone pulse therapy in Kawasaki disease patients with coronary artery aneurysms | 24 weeks from enrollment
  Measurement of body weight in Kilogram
Incidence of Treatment-Emergent Adverse Events and physical effects of Methylprednisolone pulse therapy in Kawasaki disease patients with coronary artery aneurysms | 4 weeks from enrollment
  Measurement of body height in centimeter
Incidence of Treatment-Emergent Adverse Events and physical effects of Methylprednisolone pulse therapy in Kawasaki disease patients with coronary artery aneurysms | 8 weeks from enrollment
  Measurement of body height in centimeter
Incidence of Treatment-Emergent Adverse Events and physical effects of Methylprednisolone pulse therapy in Kawasaki disease patients with coronary artery aneurysms | 12 weeks from enrollment
  Measurement of body height in centimeter
Incidence of Treatment-Emergent Adverse Events and physical effects of Methylprednisolone pulse therapy in Kawasaki disease patients with coronary artery aneurysms | 16 weeks from enrollment
  Measurement of body height in centimeter
Incidence of Treatment-Emergent Adverse Events and physical effects of Methylprednisolone pulse therapy in Kawasaki disease patients with coronary artery aneurysms | 20 weeks from enrollment
  Measurement of body height in centimeter
Incidence of Treatment-Emergent Adverse Events and physical effects of Methylprednisolone pulse therapy in Kawasaki disease patients with coronary artery aneurysms | 24 weeks from enrollment
  Measurement of body height in centimeter
Incidence of Treatment-Emergent Adverse Events and physical effects of Methylprednisolone pulse therapy in Kawasaki disease patients with coronary artery aneurysms | 4 weeks from enrollment
  Measurement of blood pressure & intraocular pressure in mmHg
Incidence of Treatment-Emergent Adverse Events and physical effects of Methylprednisolone pulse therapy in Kawasaki disease patients with coronary artery aneurysms | 8 weeks from enrollment
  Measurement of blood pressure & intraocular pressure in mmHg
Incidence of Treatment-Emergent Adverse Events and physical effects of Methylprednisolone pulse therapy in Kawasaki disease patients with coronary artery aneurysms | 12 weeks from enrollment
  Measurement of blood pressure & intraocular pressure in mmHg
Incidence of Treatment-Emergent Adverse Events and physical effects of Methylprednisolone pulse therapy in Kawasaki disease patients with coronary artery aneurysms | 16 weeks from enrollment
  Measurement of blood pressure & intraocular pressure in mmHg
Incidence of Treatment-Emergent Adverse Events and physical effects of Methylprednisolone pulse therapy in Kawasaki disease patients with coronary artery aneurysms | 20 weeks from enrollment
  Measurement of blood pressure & intraocular pressure in mmHg
Incidence of Treatment-Emergent Adverse Events and physical effects of Methylprednisolone pulse therapy in Kawasaki disease patients with coronary artery aneurysms | 24 weeks from enrollment
  Measurement of blood pressure & intraocular pressure in mmHg
Incidence of Treatment-Emergent Adverse Events and physical effects of Methylprednisolone pulse therapy in Kawasaki disease patients with coronary artery aneurysms | 4 weeks from enrollment
  Measurement of Sodium, Potassium, Chlorine level in blood in MEQ/L
Incidence of Treatment-Emergent Adverse Events and physical effects of Methylprednisolone pulse therapy in Kawasaki disease patients with coronary artery aneurysms | 8 weeks from enrollment
  Measurement of Sodium, Potassium, Chlorine level in blood in MEQ/L
Incidence of Treatment-Emergent Adverse Events and physical effects of Methylprednisolone pulse therapy in Kawasaki disease patients with coronary artery aneurysms | 12 weeks from enrollment
  Measurement of Sodium, Potassium, Chlorine level in blood in MEQ/L
Incidence of Treatment-Emergent Adverse Events and physical effects of Methylprednisolone pulse therapy in Kawasaki disease patients with coronary artery aneurysms | 16 weeks from enrollment
  Measurement of Sodium, Potassium, Chlorine level in blood in MEQ/L
Incidence of Treatment-Emergent Adverse Events and physical effects of Methylprednisolone pulse therapy in Kawasaki disease patients with coronary artery aneurysms | 20 weeks from enrollment
  Measurement of Sodium, Potassium, Chlorine level in blood in MEQ/L
Incidence of Treatment-Emergent Adverse Events and physical effects of Methylprednisolone pulse therapy in Kawasaki disease patients with coronary artery aneurysms | 24 weeks from enrollment
  Measurement of Sodium, Potassium, Chlorine level in blood in MEQ/L
Incidence of Treatment-Emergent Adverse Events and physical effects of Methylprednisolone pulse therapy in Kawasaki disease patients with coronary artery aneurysms | 4 weeks from enrollment
  Measurement of Calcium & Fibrinogen level in blood in mg/dl
Incidence of Treatment-Emergent Adverse Events and physical effects of Methylprednisolone pulse therapy in Kawasaki disease patients with coronary artery aneurysms | 8 weeks from enrollment
  Measurement of Calcium & Fibrinogen level in blood in mg/dl
Incidence of Treatment-Emergent Adverse Events and physical effects of Methylprednisolone pulse therapy in Kawasaki disease patients with coronary artery aneurysms | 12 weeks from enrollment
  Measurement of Calcium & Fibrinogen level in blood in mg/dl
Incidence of Treatment-Emergent Adverse Events and physical effects of Methylprednisolone pulse therapy in Kawasaki disease patients with coronary artery aneurysms | 16 weeks from enrollment
  Measurement of Calcium & Fibrinogen level in blood in mg/dl
Incidence of Treatment-Emergent Adverse Events and physical effects of Methylprednisolone pulse therapy in Kawasaki disease patients with coronary artery aneurysms | 20 weeks from enrollment
  Measurement of Calcium & Fibrinogen level in blood in mg/dl
Incidence of Treatment-Emergent Adverse Events and physical effects of Methylprednisolone pulse therapy in Kawasaki disease patients with coronary artery aneurysms | 24 weeks from enrollment
  Measurement of Calcium & Fibrinogen level in blood in mg/dl
Incidence of Treatment-Emergent Adverse Events and physical effects of Methylprednisolone pulse therapy in Kawasaki disease patients with coronary artery aneurysms | 4 weeks from enrollment
  Measurement of prothrombin time & activated partial thromboplastin time in second
Incidence of Treatment-Emergent Adverse Events and physical effects of Methylprednisolone pulse therapy in Kawasaki disease patients with coronary artery aneurysms | 8 weeks from enrollment
  Measurement of prothrombin time & activated partial thromboplastin time in second
Incidence of Treatment-Emergent Adverse Events and physical effects of Methylprednisolone pulse therapy in Kawasaki disease patients with coronary artery aneurysms | 12 weeks from enrollment
  Measurement of prothrombin time & activated partial thromboplastin time in second
Incidence of Treatment-Emergent Adverse Events and physical effects of Methylprednisolone pulse therapy in Kawasaki disease patients with coronary artery aneurysms | 16 weeks from enrollment
  Measurement of prothrombin time & activated partial thromboplastin time in second
Incidence of Treatment-Emergent Adverse Events and physical effects of Methylprednisolone pulse therapy in Kawasaki disease patients with coronary artery aneurysms | 20 weeks from enrollment
  Measurement of prothrombin time & activated partial thromboplastin time in second
Incidence of Treatment-Emergent Adverse Events and physical effects of Methylprednisolone pulse therapy in Kawasaki disease patients with coronary artery aneurysms | 24 weeks from enrollment
  Measurement of prothrombin time & activated partial thromboplastin time in second
Incidence of Treatment-Emergent Adverse Events and physical effects of Methylprednisolone pulse therapy in Kawasaki disease patients with coronary artery aneurysms | 4 weeks from enrollment
  Measurement of protein C & protein S level in ％
Incidence of Treatment-Emergent Adverse Events and physical effects of Methylprednisolone pulse therapy in Kawasaki disease patients with coronary artery aneurysms | 8 weeks from enrollment
  Measurement of protein C & protein S level in ％
Incidence of Treatment-Emergent Adverse Events and physical effects of Methylprednisolone pulse therapy in Kawasaki disease patients with coronary artery aneurysms | 12 weeks from enrollment
  Measurement of protein C & protein S level in ％
Incidence of Treatment-Emergent Adverse Events and physical effects of Methylprednisolone pulse therapy in Kawasaki disease patients with coronary artery aneurysms | 16 weeks from enrollment
  Measurement of protein C & protein S level in ％
Incidence of Treatment-Emergent Adverse Events and physical effects of Methylprednisolone pulse therapy in Kawasaki disease patients with coronary artery aneurysms | 20 weeks from enrollment
  Measurement of protein C & protein S level in ％
Incidence of Treatment-Emergent Adverse Events and physical effects of Methylprednisolone pulse therapy in Kawasaki disease patients with coronary artery aneurysms | 24 weeks from enrollment
  Measurement of protein C & protein S level in ％

SECONDARY OUTCOMES:
Echocardiography on the coronary artery lesion of Kawasaki disease | 4 weeks from enrollment
  Use echocardiography to measure the diameter of coronary artery (including right coronary artery [RCA], left coronary artery [LCA] and left anterior descending [LAD]) to investigate the regression of coronary artery dilatation or aneurysm formation. The dilatation is define the diameter of coronary artery. For children under 5 yrs, the diameter should not be wider than 3mm. For children over 5 yrs, the diameter should not be wider than 4mm. Adjacent segment artery should not be wider than 1.5 times.
Echocardiography on the coronary artery lesion of Kawasaki disease | 8 weeks from enrollment
  Use echocardiography to measure the diameter of coronary artery (including right coronary artery [RCA], left coronary artery [LCA] and left anterior descending [LAD]) to investigate the regression of coronary artery dilatation or aneurysm formation. The dilatation is define the diameter of coronary artery. For children under 5 yrs, the diameter should not be wider than 3mm. For children over 5 yrs, the diameter should not be wider than 4mm. Adjacent segment artery should not be wider than 1.5 times.
Echocardiography on the coronary artery lesion of Kawasaki disease | 12 weeks from enrollment
  Use echocardiography to measure the diameter of coronary artery (including right coronary artery [RCA], left coronary artery [LCA] and left anterior descending [LAD]) to investigate the regression of coronary artery dilatation or aneurysm formation. The dilatation is define the diameter of coronary artery. For children under 5 yrs, the diameter should not be wider than 3mm. For children over 5 yrs, the diameter should not be wider than 4mm. Adjacent segment artery should not be wider than 1.5 times.
Echocardiography on the coronary artery lesion of Kawasaki disease | 16 weeks from enrollment
  Use echocardiography to measure the diameter of coronary artery (including right coronary artery [RCA], left coronary artery [LCA] and left anterior descending [LAD]) to investigate the regression of coronary artery dilatation or aneurysm formation. The dilatation is define the diameter of coronary artery. For children under 5 yrs, the diameter should not be wider than 3mm. For children over 5 yrs, the diameter should not be wider than 4mm. Adjacent segment artery should not be wider than 1.5 times.
Echocardiography on the coronary artery lesion of Kawasaki disease | 20 weeks from enrollment
  Use echocardiography to measure the diameter of coronary artery (including right coronary artery [RCA], left coronary artery [LCA] and left anterior descending [LAD]) to investigate the regression of coronary artery dilatation or aneurysm formation. The dilatation is define the diameter of coronary artery. For children under 5 yrs, the diameter should not be wider than 3mm. For children over 5 yrs, the diameter should not be wider than 4mm. Adjacent segment artery should not be wider than 1.5 times.
Echocardiography on the coronary artery lesion of Kawasaki disease | 24 weeks from enrollment
  Use echocardiography to measure the diameter of coronary artery (including right coronary artery [RCA], left coronary artery [LCA] and left anterior descending [LAD]) to investigate the regression of coronary artery dilatation or aneurysm formation. The dilatation is define the diameter of coronary artery. For children under 5 yrs, the diameter should not be wider than 3mm. For children over 5 yrs, the diameter should not be wider than 4mm. Adjacent segment artery should not be wider than 1.5 times.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No